CLINICAL TRIAL: NCT03604289
Title: Cardiovascular Effects of Angiotensin 1-7 in Obesity Hypertension
Brief Title: Angiotensin 1-7 in Obesity Hypertension
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding terminated
Sponsor: Amy Arnold (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Amy Arnold, Associate Professor, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY00008170; 18POST33960087 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Obesity; Hypertension
Keywords: angiotensin-1-7
MeSH Terms: conditions — Obesity; Hypertension | interventions — angiotensin I (1-7); Acetates; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Angiotensin-(1-7) (Experimental): Participants receive intravenous angiotensin-(1-7) at one study visit for 100 minutes total. Angiotensin-(1-7) will be given in escalating doses of 2ng/kg/min, 4ng/kg/min, and 8ng/kg/min. Each of these doses will be infused for 10 minutes. Following the dose escalation, angiotensin-(1-7) will be given at 8ng/kg/min for an additional 70 minutes. Infusion rates will be calculated for each patient based on body mass.
  Interventions: Drug: Angiotensin-(1-7)
- Saline (Placebo Comparator): Participants receive intravenous saline at one study visit for 100 minutes total. The volume of saline will match the volume of angiotensin-(1-7) infused. Infusion rates will be calculated for each patient based on body mass. Saline will be given in escalating doses for 10 minutes each and then held for 70 minutes at the highest dose.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Angiotensin-(1-7) — This is a biologically active endogenous angiotensin peptide that may play an important role in regulation of blood pressure.
  Other Names: Angiotensin I/II (1-7) Acetate
  Arms: Angiotensin-(1-7)
Drug: Saline — Saline will be used as the placebo comparator
  Other Names: Normal saline; 0.9% sodium chloride
  Arms: Saline

SUMMARY:
The purpose of this study is to find out if the investigational drug angiotensin-(1-7) improves cardiovascular health in patients with obesity and high blood pressure.

DETAILED DESCRIPTION:
Obesity is a major public health concern that greatly increases risk for developing cardiovascular disease. Importantly, obesity is associated with endothelial dysfunction and elevated sympathetic tone, vascular and autonomic derangements known to elevate blood pressure and increase cardiovascular risk. The renin-angiotensin system may explain cardiovascular complications in obesity. Angiotensin-(1-7) is a beneficial hormone that is reduced in obesity and restoration of this hormone improves endothelial function and reduces sympathetic activity in animal models, which may contribute to its blood pressure-lowering effects. The investigators will test the hypothesis that angiotensin-(1-7) improves cardiovascular function in humans with obesity hypertension. This hypothesis will be tested in a randomized, double blind, placebo-controlled crossover study. The investigators will measure the effects of acute intravenous angiotensin-(1-7) infusion on endothelial-mediated vasodilation in the brachial and coronary arteries and on blood pressure and muscle sympathetic nerve activity with direct microneurography recordings in obese hypertensive humans.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all races
* Capable of giving informed consent
* Age 18-60 years
* Body mass index (BMI) between 30-40 kg/m2
* Hypertension defined as two or more seated blood pressure readings >130/80 mmHg or use of anti-hypertensive medications
* Satisfactory history and physical exam

Exclusion Criteria:

* Age ≤ 17 or ≥ 61 years
* Pregnant or nursing women
* Decisional impairment
* Prisoners
* Alcohol or drug abuse
* Current smokers
* Highly trained athletes
* Subjects with >5% weight change in the past 3 months
* Evidence of type I or type II diabetes (fasting glucose > 126 mg/dL or use of anti-diabetic medications)
* History of serious cardiovascular disease (e.g. myocardial infarction within 6 months, symptomatic coronary artery disease, presence of angina pectoris, significant arrhythmia, congestive heart failure, deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis, hypertrophic cardiomyopathy) or cerebrovascular disease (e.g. cerebral hemorrhage, stroke, transient Ischemic attack).
* History or presence of immunological or hematological disorders
* Impaired hepatic function (AST or ALT levels >2 times upper limit of normal range)
* Impaired renal function (serum creatinine >2.0 mg/dl)
* Anemia
* Treatment with serotonin-norepinephrine reuptake inhibitors (SNRIs) or norepinephrine transporter (NET) inhibitors
* Treatment with phosphodiesterase-5 inhibitors
* Treatment with anticoagulants (e.g. warfarin)
* Treatment with chronic systemic glucocorticoid therapy (>7 consecutive days in 1 month)
* Treatment with any investigational drug in the 1-month preceding the study
* Inability to give, or withdraw, informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Change in brachial artery diameter with reactive hyperemia | 15 minutes including baseline, cuff inflation, and reactive hyperemia
  A blood pressure cuff will be inflated to a suprasystolic pressure for 5 minutes then deflated. Brachial artery diameter will be measured continuously before, during, and after cuff inflation using duplex ultrasound.

SECONDARY OUTCOMES:
Heart Rate Variability | 30 minutes
  Resting heart rate variability will be calculated from baseline blood pressure recordings
Circulating catecholamines | 5 minutes
  circulating catecholamines will be measured from blood samples
Change in coronary blood velocity to the cold pressor test | 20 minutes
  Coronary blood velocity will be measured using duplex ultrasound before, during, and after cold pressor test (hand in ice water for 2 minutes)
Change in systolic and diastolic blood pressure to the cold pressor test | 20 minutes
  Blood pressure will be measured continuously with a finger cuff before, during, and after the cold pressor test.
Change in muscle sympathetic nerve activity to the cold pressor test | 20 minutes
  Muscle sympathetic nerve activity will be measured using peroneal nerve microneurography before, during, and after the cold pressor test.

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Arnold, Ph.D., Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States